CLINICAL TRIAL: NCT01705444
Title: The Impact of the Temporary Stent on Parameters of Voiding Function and on the Quality of Life Among Patients With LUTS
Brief Title: The Spanner Prostatic Stent and Patient's Quality of Life
Acronym: SpannerQoL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Princess Al-Johara Al-Ibrahim Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-11-541; E-11-541 (Other: Institutional Review Board)
Record Dates: First submitted 2012-10-09; First posted 2012-10-12 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2012-10

CONDITIONS: Prostatic Obstruction
Keywords: Urinary retention; Foley catheter; The Spanner; Quality of life
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Foley catheter and The Spanner Insertion (Other): Quality of life questionnaire after using the Foley catheter and the Spanner
  Interventions: Device: Foley Catheter and The Spanner Insertion

INTERVENTIONS:
Device: Foley Catheter and The Spanner Insertion — A Foley catheter will be inserted for 3-5 days, then a voiding trail will be attempted by the patient himself without the catheter. Then, the Spanner will be inserted into the same patient for another 3-5 days and an evacuation trail will be attempted also by the patient after removal of the Spanner. Treatment Satisfaction Questionnaire (TSQ) will be applied by the same person to the patient twice, once after removal of the Foley catheter and the second after removal of the Spanner.
  Other Names: Foley Catheter; The Spanner

SUMMARY:
Acute urinary retention is considered one of the most common problems in the older age, especially those who have benign prostatic hyperplasia. Solving the problem of acute urinary retention using the Foley catheter still causes problems at the level of patient movement and the daily exercises. However, with the emergence of a new device, the spanner, investigators believe that many of the above mentioned problems can be resolved. This tool may provide more freedom for the patient.

DETAILED DESCRIPTION:
This research comes up to date with technological innovations in the field of health where investigators want to evaluate the efficacy of a new catheter (The Spanner) to reduce the acute urinary retention and to determine whether they are consistent with the daily life of the patient, compared to the Foley catheter previously used.

The study include all patients with acute urinary retention due to prostatic obstruction. Subjects were excluded if they had prior surgery for prostate cancer, had any other urethral or bladder surgery, or if they were at high risk of developing bladder or kidney stones The study will be national community based study conducted in different hospitals in Saudi Arabia. Investigators will test two different types of stents in patients with acute urinary retention for a short period (not exceeding five days), find out the compatibility of these stents with the daily life of the patient and determine their impact on his quality of life using an appropriate questionnaire after each use.

ELIGIBILITY:
Inclusion Criteria:

* Acute Urinary retention due to Prostatic Obstruction

Exclusion Criteria:

* Subjects were excluded if they had prior surgery for prostate cancer, had any other urethral or bladder surgery, or if they were at high risk of developing bladder or kidney stones

Ages: 45 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2012-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Quality of life questionnaire after using the Foley catheter | After five days
  Using a validated Quality of life questionnaire designed for the study

SECONDARY OUTCOMES:
Quality of life questionnaire after using the spanner | After five days
  Using the same Quality of life questionnaire

OTHER OUTCOMES:
IPSS international prostate symptom score assessment | After five days of using the Spanner
  Assessment of the prostate symptom score using the IPSS questionnaire five days after using the Spanner

CONTACTS AND LOCATIONS:
Overall Officials: Danny M. Rabah, MD, Principal Investigator — Princess Al-Johara Al-Ibrahim Cancer Research Center
Locations (1):
- Princess Al-Johara Cancer Research Center, Riyadh, Saudi Arabia, Riyadh, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in per-reviewed journal